CLINICAL TRIAL: NCT02684227
Title: A Phase II Study With a Limited Safety Lead-In of Enzalutamide in Combination With Carboplatin and Paclitaxel in Advanced Stage or Recurrent Endometrioid Endometrial Cancer
Brief Title: Enzalutamide, Carboplatin, and Paclitaxel in Treating Patients With Stage III-IV or Recurrent Endometrioid Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0723; NCI-2016-00562 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0723 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Endometrial Endometrioid Adenocarcinoma; Recurrent Uterine Corpus Carcinoma; Stage III Uterine Corpus Cancer AJCC v7; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IV Uterine Corpus Cancer AJCC v7; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Uterine Corpus Cancer AJCC v7
MeSH Terms: interventions — Carboplatin; enzalutamide; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enzalutamide, paclitaxel, carboplatin) (Experimental): Patients receive enzalutamide PO QD alone on days 1-28. Patients then receive enzalutamide PO QD on days 1-21, paclitaxel IV over 3 hours on day 1, and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 6-9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Enzalutamide; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well enzalutamide, carboplatin, and paclitaxel work in treating patients with endometrioid endometrial cancer that is stage III-IV or has come back. Androgens can cause the growth of endometrioid endometrial cancer. Antihormone therapy, such as enzalutamide may lessen the amount of androgen made by the body. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving enzalutamide, carboplatin, and paclitaxel may work better in treating patients with endometrioid endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical activity of combination enzalutamide, carboplatin and paclitaxel represented as:

Ia. Objective tumor response (complete response [CR] + partial response [PR]). Ib. The proportion of patients who survive progression-free for at least 6 months after initiating therapy.

II. To quantify protein and phosphoprotein expression of androgen receptor (AR) and AR-response genes following enzalutamide treatment in match-paired pre and post treatment tumor biopsies.

III. To determine the safety and feasibility of daily enzalutamide given in combination with carboplatin and paclitaxel in women with advanced stage or recurrent endometrial cancer.

SECONDARY OBJECTIVES:

I. Determine median response duration. II. Estimate progression free survival and overall survival. III. Evaluate for presence of pharmacokinetic interaction between enzalutamide and paclitaxel.

EXPLORATORY OBJECTIVES:

I. Correlate molecular results, including AR receptor expression and activation, to clinical endpoints.

II. Identify potential agents to synergize with enzalutamide based on pathways activated after enzalutamide treatment.

OUTLINE:

Patients receive enzalutamide orally (PO) once daily (QD) alone on days 1-28. Patients then receive enzalutamide PO QD on days 1-21, paclitaxel intravenously (IV) over 3 hours on day 1, and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 6-9 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis (by either primary surgical specimen or biopsy for recurrence) of advanced stage (stage III or IV) or recurrent endometrioid endometrial cancer
* Measurable disease (at least one measurable lesion) IS required; a measurable lesion is one that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be > 10 mm when measured by computed tomography (CT) scan, magnetic resonance imaging (MRI), or caliper measurement by clinical exam; or > 20 mm when measured by chest x-ray; lymph nodes must be > 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by Response Evaluation Criteria in Solid Tumors (RECIST); tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patient with an Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy of greater than 3 months in the opinion of the principal investigator
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration
* PRIOR THERAPY: Patients should have had NO prior chemotherapy agents for advanced or recurrent endometrial cancer; prior chemotherapy administration in conjunction with primary radiation therapy as a radiosensitizer would NOT exclude a patient from participation in this trial
* Absolute neutrophil count (ANC) >= 1,500/mcl, equivalent to Common Terminology Criteria (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4.03) grade 1
* Platelets >= 100,000/mcl
* Calculated creatinine clearance (Cockcroft-Gault formula) > 50 ml/min OR 24-hour urine creatinine clearance > 50 ml/min
* Bilirubin =< 1.5 x upper limit of normal (ULN) (CTCAE v4.03 grade 1; in patients with known Gilbert syndrome, a total bilirubin =< 3.0 x ULN, with direct bilirubin =< 1.5 x ULN)
* Aspartate aminotransferase (AST) and alkaline phosphatase =< 2.5 x ULN (CTCAE v4.03 grade 1; AST and alanine aminotransferase [ALT] =< 3 x ULN [or =< 5.0 x ULN if hepatic metastases are present])
* Neuropathy (sensory and motor) =< CTCAE v4.03 grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) =< 1.5 times the institutional upper limit of normal; patients receiving low molecular weight heparin for the prevention or treatment of venous thromboembolic disease are eligible if considered clinically stable on their regimen
* Patients must have signed an approved informed consent
* Because no dosing or adverse event data are currently available on the use of enzalutamide in combination with carboplatin and paclitaxel in patients <18 years of age, children are excluded from this study.
* The effects of enzalutamide on the developing human fetus are unknown; for this reason and because therapeutic agents used in this trial may be teratogenic, women of child-bearing potential and their partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women of child-bearing potential (intact uterus) should have a negative serum pregnancy test. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must be able to swallow whole tablets
* With the exception of alopecia, any unresolved toxicities from prior chemotherapy should be no greater than CTCAE v4 grade 1 at the time of starting study treatment
* Patients on the Phase II portion only must be willing to undergo pre- and post-treatment biopsies and have at least one lesion amenable to biopsy

Exclusion Criteria:

* Patients who have isolated recurrences (vaginal, pelvic, or paraaortic) that are amenable to potentially curative treatment with radiation therapy or surgery
* Patients with the following histologies of endometrial cancer are not eligible for enrollment: papillary serous adenocarcinoma, clear cell carcinoma, adenosquamous carcinoma, mucinous adenocarcinoma, carcinosarcoma, sarcoma
* Prior Therapy:

  * Prior Chemotherapy: Patients who have had a prior chemotherapy regimen for advanced or metastatic disease are excluded
  * Prior Radiation Therapy: Patients may have received prior radiation therapy for treatment of endometrial carcinoma; prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, and/or intravaginal brachytherapy, alone or with chemotherapy as a radiation sensitizer; all radiation therapy must be completed at least 4 weeks prior to the first date of study therapy, the prior radiation field, radiation dose, number of fractions and prior radiation start and stop dates must be provided at registration
* Patients who have previously received enzalutamide; patients may have received prior hormonal therapy for treatment of endometrial carcinoma; all hormonal therapy must be discontinued at least one week prior to the first date of study therapy
* Patients who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events (CTCAE v4.03 grade 2 or greater, excluding alopecia) due to agents administered more than 4 weeks earlier
* Patients may not receive any other anti-neoplastic or investigational agents within 3 weeks of study enrollment; patients may not be receiving any other investigational agents during treatment on protocol
* Patients may not receive strong cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8) inhibitors, CYP2C8 inducers, or cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers; in addition, patients should not receive drugs that are metabolized by CYP3A4 or cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9)
* Patients who are pregnant or nursing; women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patient had major surgery within 28 days prior to starting study drug or has not recovered from major side effects of the surgery
* Patients may not have a history of other malignancies except for basal cell or squamous cell skin cancer, in situ cervical cancer, unless they have been disease-free for at least five years
* Patients with predisposing factors for seizure including history of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within the past 12 months, cerebral vascular accident, brain metastasis, and brain arteriovenous malformation
* Patient with history of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to enzalutamide, carboplatin, or paclitaxel
* Patients may not have symptomatic, uncontrolled spinal cord compression and/or brain metastases; a scan to confirm absence of brain metastasis is not required; patients can receive a stable dose of corticosteroids before/ during study if these were started at least 28 days prior to entry
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases (e.g., severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease], uncontrolled chronic renal diseases [glomerulonephritis, nephritic syndrome, Fanconi syndrome or renal tubular acidosis]), or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension (blood pressure >= 160/90), active bleeding diatheses or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus; screening for chronic conditions is not required
* As judged by the investigator, the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 08/24/2016 and closed to new patient entry on 06/07/2021. The study was completed on 09/27/2023 and all recruitment was done in a medical clinic setting.
Groups:
- Part A (Safety Lead-In): Enzalutamide 160 mg PO daily + Paclitaxel 175 mg/m2 on Day 1 + Carboplatin at AUC 5 on Day 1 of each 21 day cycle for 6-9 cycles
- Part B (Phase II): Enzalutamide 160 mg PO daily X21 days alone then Enzalutamide 160 mg PO daily + Paclitaxel 175 mg/m2 on Day 1 + Carboplatin at AUC 5 on Day 1 of each 21 day cycle for 6-9 cycles
Period: Overall Study
Arm/Group | Part A (Safety Lead-In) | Part B (Phase II)
Started | 7 | 43
Completed | 6 | 31
Not Completed | 1 | 12
Not completed — Adverse Event | 1 | 7
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progressive Disease | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (Safety Lead-In) | Part B (Phase II) | Total
Number analyzed (Participants) | 7 | 43 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 28 | 30
  >=65 years | 5 | 15 | 20
Age, Continuous [Mean (Full Range); unit: years] | 64.3 [54 to 76] | 61.5 [22 to 81] | 62.5 [22 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 43 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 5 | 37 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 37 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Activity of Combination Enzalutamide, Carboplatin and Paclitaxel Represented as Objective Tumor Response (Complete Response (CR) + Partial Response (PR)).
Description: No dose-limiting toxicities were observed during the safety lead-in. Objective tumor response (complete response (CR) + partial response (PR)).
Time Frame: up to 6.4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part A: Enzalutamide 160 mg PO daily + Paclitaxel 175 mg/m2 on Day 1 + Carboplatin at AUC 5 on Day 1 of each 21 day cycle for 6-9 cycles
- Part B: Enzalutamide 160 mg PO daily X21 days alone then Enzalutamide 160 mg PO daily + Paclitaxel 175 mg/m2 on Day 1 + Carboplatin at AUC 5 on Day 1 of each 21 day cycle for 6-9 cycles
Arm/Group | Part A | Part B
Number analyzed (Participants) | 7 | 43
percentage of participants | 68 [51 to 81] | 62 [44 to 78]

2. Primary Outcome: To Determine the Safety and Feasibility of Daily Enzalutamide Given in Combination With Carboplatin and Paclitaxel in Women With Advanced Stage or Recurrent Endometrial Cancer
Description: We will tabulate the adverse events by grade and relationship to study drug. Participants had at least 1 treatment-related adverse event.
Time Frame: up to 6.4 years
Measure: Number; unit: events
Arm/Group | Part A | Part B
Number analyzed (Participants) | 7 | 43
events
  Deaths (related & unrelated) | 0 | 2
  Reported SAE related to study agents | 3 | 3

3. Primary Outcome: Median Duration of Progression-free Survival
Time Frame: up to 6.4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A | Part B
Number analyzed (Participants) | 7 | 43
months | 14.23 [10.45 to NA] — Not Estimable. Insufficient number of participants with events. | 13.27 [9.86 to 25.49]

4. Secondary Outcome: Overall Survival
Time Frame: up to 6.4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A | Part B
Number analyzed (Participants) | 7 | 43
months | NA [NA to NA] — Not Estimable. Insufficient number of participants with events. | 36.14 [24.87 to NA] — Not Estimable. Insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: The study was activated on 08/24/2016 and the first patient was consented on 09/13/2016. The study was completed on 03/28/2023 when the last patient was taken off study and the study was terminated on 09/27/2023. Adverse events were reported from baseline until 30 days following the last dose of study treatment given.
Description: NCI CTCAE version 4.03
Arm/Group | Part A (Safety Lead-In) | Part B (Phase II)
All-Cause Mortality (participants affected / at risk) | 0/7 | 2/43
Serious Adverse Events (participants affected / at risk) | 3/7 | 3/43
Other Adverse Events (participants affected / at risk) | 7/7 | 32/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Safety Lead-In) (N=7) | Part B (Phase II) (N=43)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Safety Lead-In) (N=7) | Part B (Phase II) (N=43)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (5)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 17 (20)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (18) | 32 (83)
Anorexia (Metabolism and nutrition disorders) | 5 (7) | 8 (12)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (3)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac disorders - thrombus suspected (Cardiac disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 11 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 11 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 11 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 6 (6)
Edema limbs (General disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (23) | 22 (34)
Fever (General disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 2 (2)
General disorder-soreness (General disorders) | 0 (0) | 1 (1)
General disorder-forgetfulness (General disorders) | 0 (0) | 1 (2)
General muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Hallucinations (Psychiatric disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 10 (10)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 7 (12)
Hypertension (Vascular disorders) | 1 (4) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 15 (20)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 9 (14)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (6)
Infections and infestations - oral thrush (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Investigations - LDH increase (Investigations) | 1 (1) | 1 (1)
Investigations - creatinine decrease (Investigations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle weakness - upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (4) | 26 (30)
Nervous system disorders - restless leg syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (12) | 24 (59)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 24 (31)
Platelet count decreased (Investigations) | 3 (21) | 22 (59)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4)
Restlessness (Psychiatric disorders) | 0 (0) | 5 (5)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal itching (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 3 (3) | 1 (1)
White blood cell decreased (Investigations) | 2 (5) | 19 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT02684227/Prot_SAP_000.pdf